CLINICAL TRIAL: NCT02657850
Title: Multi-Institution Longitudinal Evaluation of Head and Neck Cancer Treatment - Related Dysphagia
Brief Title: Head and Neck Cancer Treatment Related Dysphagia
Status: Withdrawn | Type: Observational
Why Stopped: study approval lapsed
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: J1670; IRB00074509 (Other: JHM IRB)
Record Dates: First submitted 2016-01-11; First posted 2016-01-18 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Head and Neck Cancer; Dysphagia
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- control cohort - study subject self-reporting: Participants who have another cancer (not head and neck cancer) and undergoing treatment will self-report their dysphagia symptoms.
  Interventions: Other: non- head and neck self reporting
- study cohort - study subject self-reporting: Participants who have head and neck cancer and undergoing treatment will self-report their dysphagia symptoms.
  Interventions: Other: head neck self reporting
- study cohort - provider reporting: Participants who have head and neck cancer and undergoing treatment will have their dysphagia symptoms reported by the provider.
  Interventions: Other: provider reporting

INTERVENTIONS:
Other: non- head and neck self reporting — non- head and neck patient self reports dysphagia symptoms
  Groups: control cohort - study subject self-reporting
Other: head neck self reporting — head and neck patient self reports dysphagia symptoms
  Groups: study cohort - study subject self-reporting
Other: provider reporting — provider reports on head and neck cancer patients' dysphagia symptoms
  Groups: study cohort - provider reporting

SUMMARY:
Cancers located in the upper aerodigestive tract of the head and neck region present unique management challenges due to the crucial functions in this anatomic region along with its anatomic density. As such, cancers themselves and the actual treatment can affect these functions. Of these, the ability to effectively and safely transport a swallow bolus from the oral cavity to the esophagus is particularly important. This consideration has in fact been a major source of debate regarding the optimal management for head and neck cancers as both oncologic-effective and function-preserving therapies are desired. Accomplishing this therapeutic goal has been elusive and can be attributed to a lack of tools that effectively and longitudinally evaluate swallow function over the course of a treatment and in follow-up. As such, investigators surprisingly lack a clear understanding of the natural history of treatment -related swallow dysfunction (dysphagia) regardless of the treatment modality. As such, understanding the prevalence of this significant complication is in fact not well established. Understanding the true prevalence of treatment-related dysphagia is in fact critical to establish as it will help guide decisions as to whether or not treatment strategies require modification including de-intensification of treatment that is receiving considerable attention for favourable prognosis patients associated with the human papillomavirus (HPV).

To address this problem, winvestigators hypothesize that the quantitative and validated patient-reported outcome (PRO) instrument, the Sydney Swallow Questionnaire (SSQ), can be an effective tool to longitudinally measure swallow function to determine the natural history of head and neck cancer treatment-related swallow dysphagia. The SSQ is particularly well suited for longitudinal evaluation of swallow function as it quantifies various aspect of patient-perceived swallow function in contrast to other swallow PROs that measure the impact of swallow function on quality of life domains. To determine the two-year prevalence of dysphagia, investigators will employ a multi-institution prospective study design using our Oncospace® web-portal to facilitate secure prospective data curation and analysis that will include evaluations before, during and following standard of care definitive cancer treatment for a total of 36 months in the follow-up period.

DETAILED DESCRIPTION:
Cancers located in the upper aerodigestive tract of the head and neck region present unique management challenges due to the anatomic density of the region. These include (as for all cancers) effective management of all clinically evident cancer cells and sub-clinical cancer cells based on a knowledge of their anatomic location (2). For head and neck cancers, the anatomic density of this region of the body presents a significant risk for cancer therapies injuring important upper aerodigestive functions. In particular, swallowing function and its dysfunction (ie. dysphagia) can have multi-faceted consequences for the head and neck cancer patient including serious quality of life impairments (3) and the potential risk of late mortality with evidence to date suggest that aspiration lung injury may be a major cause (1, 4). In fact, functional considerations have had a profound influence on the history of head and neck cancer therapy development.

Historically, head and neck cancer management was managed surgically. Though oncologically effective, the transcervical exposure technique along with the tissues removed during the cancer extirpation led to increasing concerns about the functional impact of the therapy, especially as increasing interest in preserving function was sought by investigators and patients. As technical improvements in fractionated external beam radiotherapy (EBRT) developed in the early 1980s, investigations evaluated and demonstrated that various strategies to intensify EBRT with either concurrent chemotherapy or by altering the radiotherapy fractionation schedule (ie. twice daily treatments) improved not only local-regional tumour control rates but provided organ preservation. Studies now confirm that the improved local-regional control rates translate into improved survival rates and have led to their acceptance as standard-of-care (SOC) treatment options. While functional organ preservation was often described as a goal of these investigations, the ability to rigorously define and in fact measure organ function, especially swallow function, was often limited with successful organ preservation largely reflecting the ability to determine anatomic preservation (5). A major reason for this has been the limited spectrum of effective tools to not only measure function (especially swallow function) but that lend themselves to repeated systematic longitudinal use throughout a course of head and neck cancer treatment especially in follow-up surveillance where manifestations can go unappreciated. As a result, the true prevalence of treatment-related swallow dysfunction in head and neck cancer patients remains unknown, an observation confirmed in a recent multi-national systematic review (6). As noted by the Institute of Medicine, without the ability to measure, we cannot begin to improve upon the outcome (7).

Measuring swallow function in HNSCC remains a particularly challenge as efforts continue to strive towards the development of function preserving organ cancer therapy. It has arguably taken on a greater prominence in light of the changing epidemiology of OPSCC (8, 9) where an increasing number of OPSCC (oropharyngeal squamous cell cancer) patients have cancers associated with the human papillomavirus (HPV) that have a favourable prognosis regardless of whether surgical or non-surgical management approaches are undertaken (10). This changing epidemiology, which some have described in epidemic proportions (9), suggests that an increasing number of cancer survivors will be at risk of developing late complications especially those related to swallow function. While arguably this tenet remains to be firmly established, to do so highlights several challenges that are important to address. These include establishing an effective strategy to longitudinally measure swallow function that also reflects the cluster of other treatment-related symptoms that can affect swallow such as taste changes and xerostomia (6). It requires not only a valid tool but one that lends itself to repeat ease of use ideally within a patient's ecologic environment to minimize bias and preferably within an infrastructure that readily curates this measure for analysis.

To address this problem, investigators propose to longitudinally apply the Sydney Swallow Questionnaire (SSQ), a validated patient-reported outcome (PRO) instrument (11) that evaluates many dimensions of swallow function before, during treatment and in follow-up care of the head and neck cancer patient. The SSQ is particularly attractive as it is patient-centric and reflects their sensation of swallow-related symptoms (ie. xerostomia) which is important as the impact of sensory changes are otherwise not evaluated with other swallow metrics that are available. More significantly, the SSQ is quantitative, multi-dimensional (encompasses other swallow-related symptoms) and has discriminative power as a swallow metric. Normal population assessments have defined SSQ scores that reflect neurogenic and non-neurogenic dysphagia including cross-sectional studies in HNSCC patients. Its longitudinal application however has not been evaluated to define the natural history and prevalence of HNSCC-treatment related dysphagia. Lastly, our group has successfully validated a Chinese version of the SSQ (relevant for the inclusion of nasopharyngeal cancer patients due to the increase volume of the pharynx that is treated) and has developed an electronic version of both the original English and Chinese versions of the SSQ that is accessible through the web-portal of our Mosaiq/Oncospace® database that facilitates secure HIPAA-compliant data curation across institutions.

ELIGIBILITY:
Inclusion Criteria - Head and Neck Cancer Study Subjects:

1. Previously untreated head and neck cancer of any histology receiving treatment with curative oncologic intent regardless of the treatment modality.
2. Capable of providing informed consent.

Inclusion Criteria - Non-Head and Neck Cancer Study Subjects

1. Previously untreated cancer of any histology with no prior history of swallowing disorder and receiving radiation or concurrent chemoradiation or chemotherapy followed by radiation or concurrent chemoradiation.
2. Screening SSQ <234 prior to any cancer treatment.
3. Capable of providing informed consent.

Exclusion Criteria -

1. Potential study subjects who are unwilling or unable to be adherent to longitudinal assessment and follow-up. This will include potential study subjects who have poor performance status at the time of study enrollment evaluation.
2. Potential study subjects who have cognitive limitations / impairments that prevent a potential study subject's ability to provide self-reporting with the SSQ instrument and/or other data elements required as described in the study calendar.
3. Potential study subjects who have motor skill limitations that prevent a potential study subject's ability to provide self-reporting with the SSQ instrument and/or other data elements required as described in the study calendar.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: head and neck cancer
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Change in rate of dysphagia symptoms | 24 months
  To estimate the 24-month rate of dysphagia (SSQ >234 rate) as defined by the proportion of patients with total SSQ score greater than 234 at the end of 24 months follow up. This threshold value has previously been validated (1).

SECONDARY OUTCOMES:
Change in rate of dysphagia between non head and neck and head and neck patients | 24 months
  To compare the 24-month rates of dysphagia (SSQ >234 rate) between head and neck cancer patients and non-head and neck patients.
change in dysphagia across different patient treatments | 24 months
  To estimate the treatment specific rate of dysphagia (SSQ >234 rate). Treatment modality by surgery.
change in dysphagia across different patient treatments | 24 months
  To estimate the treatment specific rate of surgery with postoperative radiotherapy.
change in dysphagia across different patient treatments | 24 months
  To estimate the treatment specific rate of surgery with surgery with postoperative concurrent chemoradiation.
change in dysphagia across different patient treatments | 24 months
  To estimate the treatment specific rate of surgery with radiotherapy alone.
change in dysphagia across different patient treatments | 24 months
  To estimate the treatment specific rate of surgery with concurrent chemoradiation and induction chemotherapy followed by concurrent chemoradiation.
change in rate of secondary treatment side effect | 24 months
  To explore treatment effects on other secondary endpoint: pain visual analog scale
change in rate of secondary treatment side effect | 24 months
  To explore treatment effects on other secondary endpoint: speech-language pathology (SLP) recommended swallow exercise adherence status.
change in rate of secondary treatment side effect | 24 months
  To explore treatment effects on other secondary endpoint: Functional Oral Intake Scale (FOIS) Diet Level and disease status / pattern of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Quon, M.D., Principal Investigator — The SKCCC at Johns Hopkins
Locations (9):
- United States (6):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Lennox Hill Hospital, New York, New York
  - University of Washington, Seattle, Washington
- University of New South Wales - St. George Hospital, Sydney, New South Wales, Australia
- University of Toronto - Odette Cancer Center, Toronto, Ontario, Canada
- University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes